CLINICAL TRIAL: NCT07150182
Title: The Integrated Shared Decision-making Program of Critical Hemodialysis Initiation - the Effects on Decision Conflict, Decision Regret, Anxiety and Depression Among Family Members
Brief Title: Shared Decision-Making for Families in Critical Dialysis Initiation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TMU-JIRB:N202303124
Record Dates: First submitted 2025-08-24; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury; Decision Making ,Shared; Emotional Dysfunction
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): received integrated shared decision-making program
  Interventions: Other: The Integrated Shared Decision-making Program
- Control group (No Intervention)

INTERVENTIONS:
Other: The Integrated Shared Decision-making Program — The Integrated Shared Decision-making Program
  Arms: Intervention group

SUMMARY:
Background:Acute kidney injury (AKI) is a frequent and serious complication in critically ill patients, often necessitating difficult decisions about starting hemodialysis. While shared decision-making (SDM) is known to improve communication, the effectiveness of structured SDM programs specifically designed for family members in this critical context is not well-established.

Aims: The primary purpose of this study is to evaluate the effectiveness of a structured shared decision-making (SDM) program for family members of patients requiring critical hemodialysis initiation. We will assess the program's impact on the quality of the decision-making process (e.g., decision conflict, regret) and the psychological well-being (e.g., anxiety, depression) of the family members.

Methods: This study is a parallel-group, randomized controlled trial. Eligible participants (family members of patients with AKI initiating hemodialysis) will be randomly assigned to either an intervention group or a control group. The intervention group will receive a structured SDM support program, while the control group will receive standard care. Primary outcomes, including decision conflict, decision regret, anxiety, and depression, will be measured at baseline and follow-up. Data will be analyzed using the generalized estimating equation (GEE) model to compare the effectiveness between the two groups.

ELIGIBILITY:
Inclusion Criteria:

(A)Patients: (1)Age ≥ 20 years. (2)Admitted to the ICU. (3)Diagnosed with acute kidney injury (AKI) requiring urgent hemodialysis. (4)No medical disputes occurred during the current hospitalization. (B) Family members:

1. Age ≥ 20 years.
2. Mentally alert and able to communicate in Mandarin or Taiwanese.
3. Key person for the patient's admission (primary contact between patient, family, and medical team).
4. Willing to participate in the clinical trial.

Exclusion Criteria:

(A) Patients:

1. Age < 20 years.
2. End-stage kidney disease already receiving renal replacement therapy (including hemodialysis, peritoneal dialysis, or kidney transplantation). (B) Family members:

(1)Unable to comply with study procedures. (2)Rarely visiting the patient (less than once every three days). (3)History of alcohol or substance abuse, mental disorders, or cognitive impairment affecting participation.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
decision conflict | Follow-up assessments will be conducted four times: at baseline, one week, two weeks, and one month after the intervention.
  This scale is used to assess family members' decisional conflict and satisfaction when facing high-risk choices. The scale consists of 16 items, with higher scores indicating greater regret regarding the decision outcome.

SECONDARY OUTCOMES:
decision regret | Follow-up assessments will be conducted four times: at baseline, one week, two weeks, and one month after the intervention.
  This scale consists of 5 items, with higher scores indicating greater regret regarding the decision outcome. this Cronbach's α was 0.84-0.86.
the quality of doctor-patient communication | Follow-up assessments will be conducted four times: at baseline, one week, two weeks, and one month after the intervention.
  This scale is used to assess the quality of communication between family members (the patient's designated healthcare proxy for the current hospitalization) and medical staff regarding the patient's condition. The scale consists of 9 items, with higher scores indicating better communication between the family and healthcare providers.
anxiety- depression status | Follow-up assessments will be conducted four times: at baseline, one week, two weeks, and one month after the intervention.
  This scale consists of 14 items, including 7 items measuring anxiety and 7 items measuring depression. Higher scores indicate greater levels of anxiety or depression

IPD SHARING:
Plan to Share IPD: No
This study has not been completed.

REFERENCES:
- [Result] Wong SPY, McFarland LV, Liu CF, Laundry RJ, Hebert PL, O'Hare AM. Care Practices for Patients With Advanced Kidney Disease Who Forgo Maintenance Dialysis. JAMA Intern Med. 2019 Mar 1;179(3):305-313. doi: 10.1001/jamainternmed.2018.6197. PMID 30667475
- [Result] Palevsky PM, Liu KD, Brophy PD, Chawla LS, Parikh CR, Thakar CV, Tolwani AJ, Waikar SS, Weisbord SD. KDOQI US commentary on the 2012 KDIGO clinical practice guideline for acute kidney injury. Am J Kidney Dis. 2013 May;61(5):649-72. doi: 10.1053/j.ajkd.2013.02.349. Epub 2013 Mar 15. PMID 23499048
- [Result] Oprea AD, Del Rio JM, Cooter M, Green CL, Karhausen JA, Nailer P, Guinn NR, Podgoreanu MV, Stafford-Smith M, Schroder JN, Fontes ML, Kertai MD. Pre- and postoperative anemia, acute kidney injury, and mortality after coronary artery bypass grafting surgery: a retrospective observational study. Can J Anaesth. 2018 Jan;65(1):46-59. doi: 10.1007/s12630-017-0991-0. Epub 2017 Nov 2. PMID 29098634
- [Result] Kerr M, Bedford M, Matthews B, O'Donoghue D. The economic impact of acute kidney injury in England. Nephrol Dial Transplant. 2014 Jul;29(7):1362-8. doi: 10.1093/ndt/gfu016. Epub 2014 Apr 21. PMID 24753459
- [Result] Hsieh YC, Lee KC, Chen PH, Su CW, Hou MC, Lin HC. Acute kidney injury predicts mortality in cirrhotic patients with gastric variceal bleeding. J Gastroenterol Hepatol. 2017 Nov;32(11):1859-1866. doi: 10.1111/jgh.13777. PMID 28271564
- [Result] Hemmat V, Corbett C. Palliative Care for Nephrology Patients in the Intensive Care Unit. Crit Care Nurs Clin North Am. 2022 Dec;34(4):467-479. doi: 10.1016/j.cnc.2022.07.003. Epub 2022 Oct 12. PMID 36336436
- [Result] Groenwold RH. Falsification end points for observational studies. JAMA. 2013 May 1;309(17):1769-70. doi: 10.1001/jama.2013.3089. No abstract available. PMID 23632712
- [Result] Fang T, Du P, Wang Y, Chen D, Lu H, Cheng H, Hu W, Jiang D. Role Mismatch in Medical Decision-Making Participation Is Associated with Anxiety and Depression in Family Members of Patients in the Intensive Care Unit. J Trop Med. 2022 Apr 16;2022:8027422. doi: 10.1155/2022/8027422. eCollection 2022. PMID 35469334
- [Result] Chang PY, Wang HP, Chang TH, Yu JM, Lee SY. Stress, stress-related symptoms and social support among Taiwanese primary family caregivers in intensive care units. Intensive Crit Care Nurs. 2018 Dec;49:37-43. doi: 10.1016/j.iccn.2018.05.002. Epub 2018 Jun 22. PMID 29937076
- [Result] Collister D, Pannu N, Ye F, James M, Hemmelgarn B, Chui B, Manns B, Klarenbach S; Alberta Kidney Disease Network. Health Care Costs Associated with AKI. Clin J Am Soc Nephrol. 2017 Nov 7;12(11):1733-1743. doi: 10.2215/CJN.00950117. Epub 2017 Oct 19. PMID 29051143
- [Result] Becerra Perez MM, Menear M, Brehaut JC, Legare F. Extent and Predictors of Decision Regret about Health Care Decisions: A Systematic Review. Med Decis Making. 2016 Aug;36(6):777-90. doi: 10.1177/0272989X16636113. Epub 2016 Mar 14. PMID 26975351
- [Result] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Result] Bagshaw SM, Adhikari NKJ, Burns KEA, Friedrich JO, Bouchard J, Lamontagne F, McIntrye LA, Cailhier JF, Dodek P, Stelfox HT, Herridge M, Lapinsky S, Muscedere J, Barton J, Griesdale D, Soth M, Ambosta A, Lebovic G, Wald R; Canadian Critical Care Trials Group. Selection and Receipt of Kidney Replacement in Critically Ill Older Patients with AKI. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):496-505. doi: 10.2215/CJN.05530518. Epub 2019 Mar 21. PMID 30898872
- [Result] Athavale AM, Fu CY, Bokhari F, Bajani F, Hart P. Incidence of, Risk Factors for, and Mortality Associated With Severe Acute Kidney Injury After Gunshot Wound. JAMA Netw Open. 2019 Dec 2;2(12):e1917254. doi: 10.1001/jamanetworkopen.2019.17254. PMID 31825505
- [Result] Abebe A, Kumela K, Belay M, Kebede B, Wobie Y. Mortality and predictors of acute kidney injury in adults: a hospital-based prospective observational study. Sci Rep. 2021 Aug 2;11(1):15672. doi: 10.1038/s41598-021-94946-3. PMID 34341369